CLINICAL TRIAL: NCT06427668
Title: A Phase 2, Randomized, Placebo-controlled, Double-Blind Multicenter Study to Assess the Safety, Tolerability, and Pharmacodynamics (PD) in Adult Participants With Mild-to Moderate Alzheimer's Disease (AD) Administered SPG302
Brief Title: Study of SPG302 in Adult Participants With Mild-to-Moderate Alzheimer's Disease (AD)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Spinogenix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SPG302-ALZ-101
Record Dates: First submitted 2024-05-13; First posted 2024-05-24 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; synapse; neural connectivity; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Intervention Model Description: Phase 2 randomized, double-blind, placebo-controlled safety and tolerability study in adult participants with Alzheimer's Disease
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Quadruple (Participant, Care Provider, Investigator, Outcomes Assessor) Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part A: Active SPG302 to be administered to adult participants with AD (Active Comparator): Cohort 1: 12 participants with Alzheimer's Disease will be randomized in a 2:1 ratio to receive SPG302 or placebo. Study intervention will be 300 mg orally once daily for 28 days (cycle 1). All participants will receive open-label SPG302 for cycles 2-7. This arm may be expanded to cohort 2: 12 additional participants pending review of data, for additional dose exploration.
  Interventions: Drug: SPG302
- Part A: Placebo comparator to be administered to adult participants with AD (Placebo Comparator): Cohort 1: 12 participants with Alzheimer's Disease will be randomized in a 2:1 ratio to receive SPG302 or placebo. Study intervention will be placebo capsule orally daily for 28 days (cycle 1). All participants will receive open-label SPG302 for cycles 2-7. This arm may be expanded to 12 additional participants as cohort 2 pending review of data, for additional dose exploration.
  Interventions: Drug: Placebo
- Part B: Expansion Cohort (Experimental): Dose to be used and size of dosing cohort to be determined by Data Safety and Monitoring Committee following completion of Part A.
  Interventions: Drug: SPG302

INTERVENTIONS:
Drug: SPG302 — synthetic small molecule
  Arms: Part A: Active SPG302 to be administered to adult participants with AD; Part B: Expansion Cohort
Drug: Placebo — Placebo
  Arms: Part A: Placebo comparator to be administered to adult participants with AD

SUMMARY:
This phase 2 study will evaluate the safety, tolerability, clinical efficacy, pharmacokinetics, and pharmacodynamics of SPG302 in adult participants with mild-to-moderate AD.

DETAILED DESCRIPTION:
This is a phase 2, multicenter study to assess the safety, tolerability, CNS effects, pharmacokinetics, pharmacodynamics and clinical efficacy of SPG302 in adult participants with mild-to-moderate AD. The study will consist of 2 parts:

Part A: Placebo-controlled, randomized, safety and preliminary efficacy cohort with daily dosing for 28 day cycles

Part B: a randomized expansion cohort of daily dosing for 28 day cycles

ELIGIBILITY:
Inclusion Criteria:

* Age 45-85
* Diagnosis of mild to moderate AD
* Clinical laboratory values within normal range or < 1.5 times ULN
* If receiving AD-specific treatment, have been on stable dose for ≥ 3 months prior to first dose of study drug.
* Life expectancy of >2 years
* Able and willing to provide written informed consent

Exclusion Criteria:

* Any physical or psychological condition that prohibits study completion
* Known cardiac disease
* Active or history of malignancy in the past 5 years
* Serious infection that will not be resolved by first day of study intervention.
* History of clinically significant CNS event or diagnosis in the past 5 years.
* Acute illness within 30 days of Day 1
* History of suicidal behavior or suicidal ideation
* History of chronic alcohol use or substance abuse in the last 5 years
* HIV, hepatitis B and/or hepatitis C positive
* Vaccines within 14 days
* Receipt of investigational products within 30 days
* Blood donation within 30 days
* Pregnant or breastfeeding

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-07-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Electroencephalogram (EEG) at resting state and at auditory evoked P300 from baseline to endpoint | 8 months
  Electroencephalogram (EEG) will provide non-invasive measurement of brain activity. This test will be used to measure resting state cognitive activity as well as cognitive activity after auditory stimulation. Sound stimuli is 500Hz and 2000Hz.
Change in Alzheimer's Disease Assessment Scale-Cog (ADAS-COG) total score from baseline to endpoint | 8 months
  The Alzheimer's Disease Assessment Scale-Cognitive Subscale test (ADAS-Cog) measures language and memory, focusing on cognitive and non-cognitive functioning. It evaluates word recall, naming of objects, word recognition, comprehension and word finding. The ADAS-COG is scored 0-70. The higher the score the greater the impairment.
Change in Mini-Mental State Examination (MMSE) from baseline to endpoint | 8 months
  The Mini-Mental State Exam (MMSE) is a test of cognitive function. It includes tests of orientation, attention, memory, language and visual-spatial skills. The lower the score the greater the impairment.
C-SSRS (Columbia Suicide Severity Rating Scale) | 8 months
  Prospective suicidality assessment is performed using the Columbia-Suicide Severity Rating Scale (C-SSRS), a questionnaire to evaluate suicidal ideation and behavior. Answer "yes" on item 4 or 5 of the Suicidal Ideation section or "yes" on any item of the Suicidal Behavior section is considered positive. The suicidal behavior lethality sub-scale inquires about the level of actual or potential medical damage.
Change in Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS - CGIC) from baseline to endpoint | 8 months
  The Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS - CGIC) is a metric for clinical assessment of symptom severity. It consists of 2 parts. First a baseline evaluation of patient and caregiver is performed to collect necessary clinical information. The clinician will then conduct the second phase of the assessment after a specified time period, and changes in symptom severity are indicated on a seven point scale. A higher scale indicates a worsening of symptoms.
Change in Alzheimer's Disease Cooperative Study - Activities of Daily Living Scale from baseline to endpoint | 8 months
  The Alzheimer's Disease Cooperative Study - Activities of Daily Living Scale is an scale that assesses the performance of daily tasks and activities. A lower score indicates lower functional performance.
Quality of Life in Alzheimer's Disease (QOL-AD) from baseline to endpoint | 8 months
  The Quality of Life in Alzheimer's Disease (QOL-AD) is a test to evaluate the quality of life through a series of questions of ability to complete daily activities and tasks. A lower score indicates lower functional quality of life.

SECONDARY OUTCOMES:
Safety and tolerability of SPG302 | 8 months
  Incidence, nature and severity of adverse events (AEs) and serious adverse events (SAEs)
Plasma pharmacokinetics of SPG302 in participants with AD-Maximum Plasma Concentration (Cmax) | 8 months
  Blood will be collected following administration of SPG302 and plasma levels will be evaluated to measure the maximum concentration.
Change in biomarkers in participants with AD from baseline to endpoint. | 8 months
  To assess the effect of SPG302 on Neurofilament light (NfL), a protein elevated in AD. This will be measured in picometers/milliliter.

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Priest, MBBS, Principal Investigator — Flinders Medical Center, Adelaide, SA, Australia; Brew Brew, MBBS,MD,DSC, Principal Investigator — St Vincents Hospital, Sydney, NSW, Australia
Locations (2):
- Australia (2):
  - St Vincent's Hospital, Sydney, New South Wales
  - Flinders Medical center, Adelaide, South Australia